CLINICAL TRIAL: NCT06162754
Title: What do Parents Know About Space Maintainers: Its Relationship With Parents' Oral Health Literacy and Children's Oral Health
Brief Title: What do Parents Know About Space Maintainers
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sema Aydınoglu, associated professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2022/140
Record Dates: First submitted 2023-10-25; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Oral Health; Dental Caries in Children; Tooth Loss
Keywords: oral health literacy; space maintainer; dental caries
MeSH Terms: conditions — Tooth Loss; Dental Caries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A questionnaire and TREALD scales were applied to parents. — The survey, which included questions about sociodemographic characteristics and space maintainer awareness, was administered to parents face to face. Then, parents' oral health literacy levels were measured with TREALD-30 and TREALD-30A scales.

SUMMARY:
Space maintainers are frequently used to prevent malocclusion problems in early primary tooth loss. Oral health literacy is defined as the capacity of individuals to learn, understand and evaluate basic oral health information. It is considered that parents' awareness of space maintainers may be affected by various factors such as their demographic characteristics and oral health literacy. The aim was to evaluate the relationship between variables by determining parents' awareness of space maintainers and their oral health literacy.

DETAILED DESCRIPTION:
This cross-sectional study included 600 children and their parents. The survey, which included questions about sociodemographic characteristics and space maintainer awareness, was administered to parents face to face. Then, parents' oral health literacy levels were measured with TREALD-30 and TREALD-30A scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients who did not require urgent treatment,
* Who did not use medication for psychiatric reasons,
* Who did not have any mental illness were included.

Exclusion Criteria:

* Those who did not meet the inclusion criteria were excluded from the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: children who applied for the dental trearment to the Faculty of Dentistry in Rize
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
the knowledge about space maintainers of the parents | for three months from the beginning of the study
  15 questions that evaluates the awareness about space maintainers of parents was applied face to face.
oral health literacy of the parents | for three months from the beginning of the study
  Oral health literacy of parents was assessed using the Turkish Rapid Estimate of Adult Literacy in Dentistry (TREALD-30 ) scale.
oral health literacy of the parents assessed by TREALD-30A scale | for three months from the beginning of the study
  Oral health literacy of parents was assessed using the Turkish Rapid Estimate of Adult Literacy in Dentistry (TREALD-30A) scale.

SECONDARY OUTCOMES:
the correlation between oral health literacy and knowledge about space maintainers of parents | for three months from the beginning of the study
  the correlation between oral health literacy and knowledge about space maintainers of parents was assessed using TREALD scales and a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sema AYDINOGLU, Principal Investigator — Recep Tayyip Erdogan University Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Recep Tayyip Erdogan University Training and Research Hospital, Rize
  - Sema AYDINOGLU, Rize